CLINICAL TRIAL: NCT03782935
Title: Early Identification of Affected Children and Nutritional Risk Factors for FASD in Ukraine
Brief Title: Nutritional Risk Factors for FASD in Ukraine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH); Omni-Net Ukraine (Unknown)
Responsible Party: Principal Investigator, Christina Chambers, Professor of Pediatrics, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 080035
Record Dates: First submitted 2018-12-18; First posted 2018-12-20 (Actual); Last update posted 2018-12-20 (Actual); Status verified 2018-12

CONDITIONS: Fetal Alcohol Spectrum Disorders
Keywords: alcohol; pregnancy; infant
MeSH Terms: conditions — Fetal Alcohol Spectrum Disorders

STUDY DESIGN:
Intervention Model Description: Pregnant women assigned to 1) over-the-counter approved prenatal multivitamin mineral supplement alone provided by the study at time of enrollment, 2)over-the-counter approved prenatal multivitamin mineral supplement with additional over-the-counter approved 750 mg choline supplement provided by the study at the time of enrollment, or 3) standard of care which is recommendation to take over-the-counter prenatal multivitamin mineral supplements
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- prenatal multivitamin mineral supplement (Experimental): received prenatal multivitamin mineral supplement at time of enrollment TheraVit multivitamin/mineral prenatal supplement with instructions to take 1 per day through the remainder of pregnancy
  Interventions: Dietary Supplement: Prenatal multivitamin mineral supplement
- prenatal multivitamin mineral supplement plus choline (Experimental): received prenatal multivitamin mineral supplement plus additional choline supplemental vitamin TheraVit multivitamin mineral supplement plus 750 mg. choline with instructions to take1 multivitamin mineral supplement and 750 mg. per day of choline through the remainder of pregnancy
  Interventions: Dietary Supplement: Prenatal multivitamin mineral supplement
- Comparison (No Intervention): Advised to follow obstetrics standard of care which is to take a prenatal vitamin/mineral supplement

INTERVENTIONS:
Dietary Supplement: Prenatal multivitamin mineral supplement — prenatal vitamin/mineral supplement with or without choline supplement
  Other Names: Prenatal multivitamin mineral supplement plus choline supplement
  Arms: prenatal multivitamin mineral supplement; prenatal multivitamin mineral supplement plus choline

SUMMARY:
Interventional study randomizing pregnant women at two sites in Ukraine who have or have not already consumed moderate to heavy levels of alcohol in pregnancy to receiving a standard prenatal vitamin supplement with or without additional choline supplement or standard of care (recommendation to take vitamin supplements) through the remainder of pregnancy, and to compare neurobehavioral performance of the offspring on the Bayley Scales of Infant Development at 12 months of age between groups. The overall sample size target was 300 alcohol exposed and 300 low or unexposed across both sites.

DETAILED DESCRIPTION:
Pregnant women coming in for routine prenatal diagnostic testing or prenatal care at two sites in Ukraine, Rivne Diagnostic Center or Khmelnytsky Regional Perinatal Center, were screened for alcohol consumption during pregnancy. Those who met the criteria of consuming 4-5 drinks per occasion on 3-4 occasions in either the month around conception or the most recent month of pregnancy were eligible for recruitment into the alcohol exposed group, and the next available woman who consumed no more than 2 drinks on any occasion in the month around conception or the most recent month of pregnancy was eligible for recruitment into the alcohol low or no exposure group. Within alcohol group and within site, women were randomized on a 1:1 basis to receiving a study-provided prenatal vitamin (TheraVit) manufactured in the U.S. and registered in Ukraine as an over-the-counter product, or to receiving standard of care which is obstetric advice to take prenatal vitamins on their own. Within the group randomized to receiving the prenatal vitamins, women were further randomized on a 1:1 basis to receiving an additional 750 mg. of supplemental choline manufactured in the U.S., and registered in Ukraine as an over-the-counter product.

Women in both cohorts were followed until delivery and those with live born children were followed until the child reached one year of age. The primary endpoint for the intervention was performance on the mental developmental index (MDI) and the psychomotor developmental index (PDI) components of the Bayley Scales of Infant Development II. The Bayley tests were administered at approximately 12 months adjusted chronological age by trained psychologists in Ukraine.

The primary comparison for the study was within the alcohol-exposed group, comparing mean Bayley scores on MDI and separately on PDI between those randomized to receiving the study prenatal vitamin and those randomized to standard of care.

Secondary comparisons for the study examined

1. the mean MDI and PDI scores on the Bayley within the alcohol-exposed group in those randomized to receiving the prenatal vitamin plus choline vs. those who received the prenatal vitamin alone
2. the mean MDI and PDI scores on the Bayley within the low or unexposed group in those who received the prenatal vitamin vs. those who did not
3. the mean MDI and PDI scores on the Bayley within the low or unexposed group in those who received the prenatal vitamin plus choline vs. those who received the prenatal vitamin alone
4. adjusted comparisons for all of the above taking into account participants who were taking vitamins on their own at the time of enrollment, and/or who were taking vitamins on their own if assigned to the standard of care group.

ELIGIBILITY:
Inclusion Criteria:

* currently pregnant
* reported alcohol consumption 4-5 drinks per occasion on 3-4 occasions in the month around conception or the most recent month of pregnancy, or
* no more than 2 drinks per occasion in either the month around conception or the most recent month of pregnancy

Exclusion Criteria:

* unable to provide consent
* unable to provide information about alcohol consumption

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 600 (Actual)
Dates: Start 2006-06; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Bayley Scales of Infant Development II Mental Developmental Index | approximately 12 months of age adjusted for preterm delivery
  Scaled score range 50 to 150 with higher scores indicating better performance
Bayley Scales of Infant Development III Psychomotor Developmental Index | approximately 12 months of age adjusted for preterm delivery
  Scaled score range 50 to 150 with higher scores indicating better performance

IPD SHARING:
Plan to Share IPD: Yes
This study is part of a collaborative initiative on Fetal Alcohol Spectrum Disorders and de-identified data is available to share with other researchers on a specified timetable with appropriate application for use.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 2020 and indefinitely
Access Criteria: Application to Collaborative Initiative on Fetal Alcohol Spectrum Disorders data oversight group at CIFASD.org
URL: http://cifasd.org